CLINICAL TRIAL: NCT03608566
Title: The Russian Registry of Patients With Severe Asthma to Collect Anonymous Long-term Evidence
Brief Title: Russian Severe Asthma Registry
Acronym: RSAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Interregional Public Organization, Russian Respiratory Society (Other)
Collaborators: AstraZeneca (Industry); Limited Liability Company Regional United System of Medical Informatization (Unknown)
Responsible Party: Sponsor
Other Study IDs: ESR-17-13479
Record Dates: First submitted 2018-05-04; First posted 2018-08-01 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-07

CONDITIONS: Severe Asthma
Keywords: severe asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Russian Severe Asthma Registry is a Russian initiative to collect anonymous long-term evidence for patients with severe asthma in Russia

DETAILED DESCRIPTION:
The Russian Severe Asthma Registry is a Russian initiative to collect anonymous long-term evidence for patients with severe asthma in Russia. The RSAR initiative is realized under the efforts of the Interregional Public Organization "Russian Respiratory Society" and LLC "RSMI" with the sponsorship of "AstraZeneca Pharmaceuticals" LLC.

The developed RSAR electronic database is a Russian software product that meets the current requirements of the Russian legislation in the field of working with personal data and the implementation of similar observational studies.

Participating researchers also agree to grant access and share anonymous data at the patient level as part of the work to implement the RSAR initiative. Participants will provide high-quality data for the development of data sets for research, approved by the Russian Respiratory Society (RPO), which has priority in owning and implementation in scientific field of the gained data. Based on ethical, legal and regulatory authorizations, anonymous data will be collected in the Central Database (CDB) on respiratory diseases (referred to here as the RSAR database) to create sets of important data and the necessary analysis. CDB is part of the software "Medical online platform ROSMED.INFO".

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years or older.

  * Patients with confirmed diagnosis of severe asthma.
  * Patients receiving treatment according to GINA step 5 or uncontrolled for 4 step. Uncontrolled patients are defined as having symptoms of severe asthma or frequent exacerbations .
  * Signed informed consent.

Exclusion Criteria:

* Patients currently participating in clinical trials at the time of enrolment

  * Intermittent, mild, moderate BA, before verification of the diagnosis.
  * COPD.
  * Diseases of the respiratory system, such as tuberculosis, sarcoidosis, IPF, lung cancer.
  * Vasculitis, systemic connective tissue diseases.
  * Neoplasm.
  * Written refusal of the patient to participate in the study after signing an informed consent.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving step 4 and 5 treatment (according to GINA, 2017) in accordance with the uncontrolled asthma severity (J.45) in health facilities
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2018-03-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
• Percentage of patients with severe asthma according frequency of exacerbations at the time of study enrollment | 03.2018 till 11.2022.
  Percentage of patients with severe asthma according frequency of exacerbations (1, 2, ≥3 exacerbations) at the time of study enrollment

SECONDARY OUTCOMES:
• Percentage of patients with severe asthma according frequency of exacerbations at the 1 year of follow-up; | 03.2019 till 11.2022.
  • Percentage of patients with severe asthma according frequency of exacerbations (1, 2, ≥3 exacerbations) at the 1 year of follow-up;
Percentage of patients with severe asthma according frequency of exacerbations at the 2 year of follow-up; | 03.2020 till 11.2022.
  • Percentage of patients with severe asthma according frequency of exacerbations (1, 2, ≥3 exacerbations) at the 2 year of follow-up;
• Percentage of patients with severe asthma according frequency of exacerbations at the 3 year of follow-up; | 03.2021 till 11.2022.
  • • Percentage of patients with severe asthma according frequency of exacerbations (1, 2, ≥3 exacerbations) at the 3 year of follow-up;
• Percentage of patients with severe asthma according frequency of exacerbations (1, 2, ≥3 exacerbations) at the 4 year of follow-up; | 03.2022 till 11.2022.
  • Percentage of patients with severe asthma according frequency of exacerbations (1, 2, ≥3 exacerbations) at the 4 year of follow-up;
• Percentage of patients with severe asthma according concomitant diseases at the time of study enrollment | 03.2018 till 11.2022.
  • Percentage of patients with severe asthma according concomitant diseases (number of observations, the mean value, the standard deviation) at the time of study enrollment
• Percentage of patients with severe asthma according concomitant diseases at the 1year of follow-up; | 03.2019 till 11.2022.
  • Percentage of patients with severe asthma according concomitant diseases (number of observations, the mean value, the standard deviation) at the 1year of follow-up;
• Percentage of patients with severe asthma according concomitant diseases at the 2 year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma according concomitant diseases (number of observations, the mean value, the standard deviation) at the 2 year of follow-up;
• Percentage of patients with severe asthma according concomitant diseases at the 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma according concomitant diseases (number of observations, the mean value, the standard deviation) at the 3 year of follow-up;
• Percentage of patients with severe asthma according concomitant diseases at the 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma according concomitant diseases (number of observations, the mean value, the standard deviation) at the 3 year of follow-up;
• • Percentage of patients with severe asthma according to parameters: age at the time of study enrollment; | 03.2018 till 11.2022
  • • Percentage of patients with severe asthma according to parameters: age (the mean value, the standard deviation) at the time of study enrollment;
• • Percentage of patients with severe asthma according to parameters: sex at the time of study enrollment; | 03.2018 till 11.2022
  • • Percentage of patients with severe asthma according to parameters: sex at the time of study enrollment;
• Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) at the time of enrollment | 03.2018 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) (the mean value, the standard deviation, the minimum value, median, maximum value) at the time of enrollment
• Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) at the 1year of follow-up; | 03.2019 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) (the mean value, the standard deviation, the minimum value, median, maximum value) at the 1year of follow-up;
• Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) at the 2year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) (the mean value, the standard deviation, the minimum value, median, maximum value) at the 2year of follow-up;
• Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) at the 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) (the mean value, the standard deviation, the minimum value, median, maximum value) at the 3year of follow-up;
• Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) at the 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of parameters: IgE (IU/ml) (the mean value, the standard deviation, the minimum value, median, maximum value) at the 4 year of follow-up;
• Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count at the time of enrollment; | 03.2018 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count (number of observations, the mean value, the standard deviation, the minimum value, median, maximum value) at the time of enrollment;
• Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count at the 1 year of follow-up; | 03.2019 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count (number of observations, the mean value, the standard deviation, the minimum value, median, maximum value) at the 1 year of follow-up;
• Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count at the 2 year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count (number of observations, the mean value, the standard deviation, the minimum value, median, maximum value) at the 2 year of follow-up;
• Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count at the 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count (number of observations, the mean value, the standard deviation, the minimum value, median, maximum value) at the 3 year of follow-up;
• Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count at the 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma with different phenotypes in terms of eosinophil levels in absolute values in complete blood count (number of observations, the mean value, the standard deviation, the minimum value, median, maximum value) at the 4 year of follow-up;
• The parameters of body mass index in the patients with severe asthma at the time of study enrollment; | 03.2018 till 11.2022
  • The parameters of body mass index (kg/m2) in the patients with severe asthma at the time of study enrollment the mean value, the standard deviation, the minimum value, median, maximum value)
• Percentage of patients with severe asthma in the parameters: of smoking at the time of study enrollment; | 03.2018 till 11.2022
  • Percentage of patients with severe asthma in the parameters: of smoking (smoker's index (pack-years)) at the time of study enrollment;
• Percentage of patients with severe asthma in the parameters: of professional history at the time of study enrollment; | 03.2018 till 11.2022
  • Percentage of patients with severe asthma in the parameters: of professional history (having or not occupational hazards at any time of life) at the time of study enrollment;
• Percentage of patients with severe asthma in the parameters: of family history at the time of study enrollment; | 03.2018 till 11.2022
  • Percentage of patients with severe asthma in the parameters: of family history at the time of study enrollment; having or not first degree relatives with asthma
• Parameters of FEV1 (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the time of study enrollment; | 03.2018 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the time of study enrollment;
• Parameters of FVC (liters, percentage of predicted)before bronchodilator in patients with severe asthma at the time of study enrollment | 03.2018 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the time of study enrollment
• Parameters of FEV1 (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the time of study enrollment; | 03.2018 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the time of study enrollment;
• Parameters of FVC (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the time of study enrollment; | 03.2018 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the time of study enrollment;
• Parameters of FEV1 (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 1 year of follow-up | 03.2019 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 1 year of follow-up
• Parameters of FVC (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 1year of follow-up; | 03.2019 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 1year of follow-up;
• Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 1 year of follow-up; | 03.2019 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 1 year of follow-up;
• Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 1year of follow-up; | 03.2019 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 1year of follow-up;
• Parameters of FEV1 (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 2 year of follow-up; | 03.2020 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 2 year of follow-up;
• Parameters of FVC (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 2year of follow-up; | 03.2020 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 2year of follow-up;
• Parameters of FEV1 (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 2 year of follow-up; | 03.2020 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 2 year of follow-up;
• Parameters of FVC (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 2year of follow-up; | 03.2020 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 2year of follow-up;
• Parameters of FEV1 (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 3 year of follow-up | 03.2021 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 3 year of follow-up
• Parameters of FVC (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 3year of follow-up | 03.2021 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 3year of follow-up
• Parameters of FEV1 (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 3 year of follow-up | 03.2021 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 3 year of follow-up
• Parameters of FVC (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 3year of follow-up | 03.2021 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 3year of follow-up
• Parameters of FEV1 (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 4 year of follow-up | 03.2022 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 4 year of follow-up
• Parameters of FVC (liters, percentage of predicted) before bronchodilator in patients with severe asthma at the 4 year of follow-up | 03.2022 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) before bronchodilator in patients with severe asthma at the 4 year of follow-up
• Parameters of FEV1 (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 4 year of follow-up; | 03.2022 till 11.2022
  • Parameters of FEV1 (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 4 year of follow-up;
• Parameters of FVC (liters, percentage of predicted) post bronchodilator in patients with severe asthma at the 4 year of follow-up; | 03.2022 till 11.2022
  • Parameters of FVC (liters, percentage of predicted) (the mean value, the standard deviation) post bronchodilator in patients with severe asthma at the 4 year of follow-up;
• Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the time of study enrollment; | 03.2018 till 11.2022
  • Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the time of study enrollment (medians, percentilies); THE ASTHMA CONTROL QUESTIONNAIRE (ACQ) The ACQ has 6 questions. In questions 1-6, patients recall their experiences during the previous 7 days and respond using a 6-point scale (0=totally controlled to 6=extremely poorly controlled).
  INTERPRETING ACQ SCORES Patients with a score of 0.75 or lower have adequately controlled asthma. Between 0.75 and 1.5 is a grey area where patients are on the borderline of adequate control. Scores over 1.5 are a strong indication of inadequate control. If a patient's score increases or decreases by greater than 0.5 between assessments, the change can be considered clinically important (justifying a change in treatment).
  SHORT-ACTING β2 AGONIST (SABA) USE NOT AVAILABLE If patients do not use a SABA, question 6 may be omitted and the mean score calculated using questions 1-5 (total score / 5).
• Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 1 year of follow-up; | 03.2019 till 11.2022
  Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 1 year of follow-up (medians, percentilies); THE ASTHMA CONTROL QUESTIONNAIRE (ACQ) The ACQ has 6 questions. In questions 1-6, patients recall their experiences during the previous 7 days and respond using a 6-point scale (0=totally controlled to 6=extremely poorly controlled).
  INTERPRETING ACQ SCORES Patients with a score of 0.75 or lower have adequately controlled asthma. Between 0.75 and 1.5 is a grey area where patients are on the borderline of adequate control. Scores over 1.5 are a strong indication of inadequate control. If a patient's score increases or decreases by greater than 0.5 between assessments, the change can be considered clinically important (justifying a change in treatment).
  SHORT-ACTING β2 AGONIST (SABA) USE NOT AVAILABLE If patients do not use a SABA, question 6 may be omitted and the mean score calculated using questions 1-5 (total score / 5).
• Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 2 year of follow-up; | 03.2020 till 11.2022
  Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 2 year of follow-up (medians, percentilies); THE ASTHMA CONTROL QUESTIONNAIRE (ACQ) The ACQ has 6 questions. In questions 1-6, patients recall their experiences during the previous 7 days and respond using a 6-point scale (0=totally controlled to 6=extremely poorly controlled).
  INTERPRETING ACQ SCORES Patients with a score of 0.75 or lower have adequately controlled asthma. Between 0.75 and 1.5 is a grey area where patients are on the borderline of adequate control. Scores over 1.5 are a strong indication of inadequate control. If a patient's score increases or decreases by greater than 0.5 between assessments, the change can be considered clinically important (justifying a change in treatment).
  SHORT-ACTING β2 AGONIST (SABA) USE NOT AVAILABLE If patients do not use a SABA, question 6 may be omitted and the mean score calculated using questions 1-5 (total score / 5).
• Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 3 year of follow-up; | 03.2021 till 11.2022
  Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 3 year of follow-up (medians, percentilies); THE ASTHMA CONTROL QUESTIONNAIRE (ACQ) The ACQ has 6 questions. In questions 1-6, patients recall their experiences during the previous 7 days and respond using a 6-point scale (0=totally controlled to 6=extremely poorly controlled).
  INTERPRETING ACQ SCORES Patients with a score of 0.75 or lower have adequately controlled asthma. Between 0.75 and 1.5 is a grey area where patients are on the borderline of adequate control. Scores over 1.5 are a strong indication of inadequate control. If a patient's score increases or decreases by greater than 0.5 between assessments, the change can be considered clinically important (justifying a change in treatment).
  SHORT-ACTING β2 AGONIST (SABA) USE NOT AVAILABLE If patients do not use a SABA, question 6 may be omitted and the mean score calculated using questions 1-5 (total score / 5).
• Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 4 year of follow-up; | 03.2022 till 11.2022
  Parameters of the analysis of the questionnaire ACQ-6 in patients with severe asthma at the 4 year of follow-up (medians, percentilies); THE ASTHMA CONTROL QUESTIONNAIRE (ACQ) The ACQ has 6 questions. In questions 1-6, patients recall their experiences during the previous 7 days and respond using a 6-point scale (0=totally controlled to 6=extremely poorly controlled).
  INTERPRETING ACQ SCORES Patients with a score of 0.75 or lower have adequately controlled asthma. Between 0.75 and 1.5 is a grey area where patients are on the borderline of adequate control. Scores over 1.5 are a strong indication of inadequate control. If a patient's score increases or decreases by greater than 0.5 between assessments, the change can be considered clinically important (justifying a change in treatment).
  SHORT-ACTING β2 AGONIST (SABA) USE NOT AVAILABLE If patients do not use a SABA, question 6 may be omitted and the mean score calculated using questions 1-5 (total score / 5).
• Number of exacerbations requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the time of study enrollment; | 03.2018 till 11.2022
  • Number of exacerbations (the mean value, the standard deviation) requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the time of study enrollment;
• Number of exacerbations requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 1year of follow-up; | 03.2019 till 11.2022
  Number of exacerbations (the mean value, the standard deviation) requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 1year of follow-up;
• Number of exacerbations requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 2year of follow-up; | 03.2020 till 11.2022
  Number of exacerbations (the mean value, the standard deviation) requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 2year of follow-up;
• Number of exacerbations requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 3 year of follow-up; | 03.2021 till 11.2022
  Number of exacerbations (the mean value, the standard deviation) requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 3 year of follow-up;
• Number of exacerbations requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 4 year of follow-up; | 03.2022 till 11.2022
  Number of exacerbations (the mean value, the standard deviation) requiring medical attention (outpatient prescription of systemic corticosteroids) in patients with severe asthma at the 4 year of follow-up;
• Number of hospitalizations in patients with severe asthma at the time of inclusion in the study; | 03.2018 till 11.2022
  • Number of hospitalizations (the mean value, the standard deviation) in patients with severe asthma at the time of inclusion in the study;
• Number of hospitalizations in patients with severe asthma at the time of inclusion in the 1 year of follow-up; | 03.2019 till 11.2022
  • Number of hospitalizations (the mean value, the standard deviation) in patients with severe asthma at the time of inclusion in the 1 year of follow-up;
• Number of hospitalizations in patients with severe asthma at the time of inclusion in the 2 year of follow-up; | 03.2020 till 11.2022
  • Number of hospitalizations (the mean value, the standard deviation) in patients with severe asthma at the time of inclusion in the 2 year of follow-up;
• Number of hospitalizations in patients with severe asthma at the time of inclusion in the 3 year of follow-up; | 03.2021 till 11.2022
  • Number of hospitalizations (the mean value, the standard deviation) in patients with severe asthma at the time of inclusion in the 3 year of follow-up;
• Number of hospitalizations in patients with severe asthma at the time of inclusion in the 4 year of follow-up; | 03.2022 till 11.2022
  • Number of hospitalizations (the mean value, the standard deviation) in patients with severe asthma at the time of inclusion in the 4 year of follow-up;
• Percentage of patients with severe asthma taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the time of study enrollment; | 03.2018 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the time of study enrollment;
• Percentage of patients with severe asthma taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 1 year of follow-up; | 03.2019 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 1 year of follow-up;
• Percentage of patients with severe asthma taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 2 year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 2 year of follow-up;
• Percentage of patients with severe asthma taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 3 year of follow-up;
• Percentage of patients with severe asthma taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking high doses of ICS/LABA, ICS/LABA+LAMA as maintenance therapy, biologics at the 4 year of follow-up;
• Percentage of patients with severe asthma taking OCS as a maintenance therapy at the time of study enrollment; | 03.2018 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking OCS as a maintenance therapy at the time of study enrollment;
• Percentage of patients with severe asthma taking OCS as a maintenance therapy at the 1 year of follow-up; | 03.2019 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking OCS as a maintenance therapy at the 1 year of follow-up;
• Percentage of patients with severe asthma taking OCS as a maintenance therapy at the 2 year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking OCS as a maintenance therapy at the 2 year of follow-up;
• Percentage of patients with severe asthma taking OCS as a maintenance therapy at the 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking OCS as a maintenance therapy at the 3 year of follow-up;
• Percentage of patients with severe asthma taking OCS as a maintenance therapy at the 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) taking OCS as a maintenance therapy at the 4 year of follow-up;
• Percentage of patients with severe asthma who have been changed therapy to 1 year of follow-up; | 03.2019 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) who have been changed therapy (step up, step down by GINA) to 1 year of follow-up;
• Percentage of patients with severe asthma who have been changed therapy to 2 year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) who have been changed therapy (step up, step down by GINA) to 2 year of follow-up;
• Percentage of patients with severe asthma who have been changed therapy to 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) who have been changed therapy (step up, step down by GINA) to 3 year of follow-up;
• Percentage of patients with severe asthma who have been changed therapy to 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma (the mean value, the standard deviation) who have been changed therapy (step up, step down by GINA) to 4 year of follow-up;
• Percentage of patients with severe asthma who called for emergency medical care for asthma at the 1 year of follow-up; | 03.2019 till 11.2022
  • Percentage of patients with severe asthma who called for emergency medical care for asthma (number of observations, the mean value, the standard deviation, median) at the 1 year of follow-up;
• Percentage of patients with severe asthma who called for emergency medical care for asthma at the 2 year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma who called for emergency medical care for asthma (number of observations, the mean value, the standard deviation, median) at the 2 year of follow-up;
• Percentage of patients with severe asthma who called for emergency medical care for asthma at the 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma who called for emergency medical care for asthma (number of observations, the mean value, the standard deviation, median) at the 3 year of follow-up;
• Percentage of patients with severe asthma who called for emergency medical care for asthma at the 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma who called for emergency medical care for asthma (number of observations, the mean value, the standard deviation, median) at the 4 year of follow-up;
• Percentage of patients with severe asthma who had disability sheets for asthma at the 1year of follow-up; | 03.2019 till 11.2022
  • Percentage of patients with severe asthma who had disability sheets for asthma (number of observations, the mean value, the standard deviation, median) at the 1year of follow-up;
• Percentage of patients with severe asthma who had disability sheets for asthma at the 2 year of follow-up; | 03.2020 till 11.2022
  • Percentage of patients with severe asthma who had disability sheets for asthma (number of observations, the mean value, the standard deviation, median) at the 2 year of follow-up;
• Percentage of patients with severe asthma who had disability sheets for asthma at the 3 year of follow-up; | 03.2021 till 11.2022
  • Percentage of patients with severe asthma who had disability sheets for asthma (number of observations, the mean value, the standard deviation, median) at the 3 year of follow-up;
• Percentage of patients with severe asthma who had disability sheets for asthma at the 4 year of follow-up; | 03.2022 till 11.2022
  • Percentage of patients with severe asthma who had disability sheets for asthma (number of observations, the mean value, the standard deviation, median) at the 4 year of follow-up;

CONTACTS AND LOCATIONS:
Overall Officials: Andrey S Belevskiy, Ph.D., Study Chair — Russian Respiratory Society
Locations (1):
- City hospital 52, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03608566/Prot_SAP_000.pdf